CLINICAL TRIAL: NCT04405102
Title: A Randomized Trial on Efficacy and Safety of Ozanimod for the Treatment of COVID-19 Patients Requiring Oxygen Support - A Pilot Trial
Brief Title: COVID-19 Ozanimod Intervention Study
Acronym: COZI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Screening was stopped by the Sponsor (43/48 participants enrolled), given the very low number of eligible patients (high vaccination rate and occurrence of the Omicron variant). The last patient randomized performed his follow-up visit.
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Collaborators: Celgene (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, François Lellouche, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-3474
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: S1P1 ligand; SARS-CoV-2; Oxygen requirement; WHO-adapted 6-points ordinal scale
MeSH Terms: conditions — COVID-19 | interventions — ozanimod; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ozanimod + standard of care (Experimental): During hospitalization, the experiment treatment of Ozanimod will be given with the standard of care (Recommendations for standard of care management of COVID-19 will be provided for anticoagulation, fluid resuscitation, corticoids and other immunomodulators, antipyretics agents, antiviral agents and other treatments. These recommendations are subject to modifications based on the new literature data.).
  Interventions: Drug: Ozanimod; Other: Standard of care
- Standard of care (Active Comparator): During hospitalization, patient will be given standard of care (Recommendations for standard of care management of COVID-19 will be provided for anticoagulation, fluid resuscitation, corticoids and other immunomodulators, antipyretics agents, antiviral agents and other treatments. These recommendations are subject to modifications based on the new literature data).
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Ozanimod — The investigational medical product (IMP) for this study is ozanimod. Ozanimod 0.23 mg be administered once daily for 4 days and then ozanimod 0.46 mg will be administered once daily for ten days.
  Other Names: Zeposia (USA)
  Arms: Ozanimod + standard of care
Other: Standard of care — During hospitalization, patient will be given standard of care (Recommendations for standard of care management of COVID-19 will be provided for anticoagulation, fluid resuscitation, corticoids and other immunomodulators, antipyretics agents, antiviral agents and other treatments. These recommendations are subject to modifications based on the new literature data).

SUMMARY:
The virus SARS-CoV-2 causes severe pneumonia which, in a proportion of patients progresses towards an Acute Respiratory Distress Syndrome (ARDS) mainly related to the antiviral immune response. To date, there is no available treatment that significantly improves outcome of patients with COVID-19 pneumonia. Sphingosine-1-phosphate receptor 1 (S1P1) ligands control vascular leakage in the airways and sphingosine-1-phosphate (S1P) receptor ligands devoid of activity on sphingosine-1-phosphate receptor 3 (S1P3) show an excellent safety profile, including ozanimod. Critically, S1P1 ligands mildly impact, but do not compromise viral clearance and they reduced lung injury in preclinical models, even without concomitant use of antivirals and with a synergistic effect when associated to antiviral agents. Ozanimod was approved by the FDA for the treatment of relapsing multiple sclerosis at the end of March 2020, and was recently (October 2020) approved by Health Canada for the same indication. The investigators believe that this immune modulator is at the top of the list of agents that should be trialed in order to mitigate the morbidity and mortality of COVID-19.

The primary objective is to substantiate the impact of ozanimod on key outcomes of COVID-19 patient progression, which will guide decision making around sample size and the choice of endpoints for future clinical trial.

ELIGIBILITY:
Inclusion criteria

* Confirmed COVID-19 (positive polymerase chain reaction (PCR) for COVID-19 from any specimen)
* Patients older than 18 years old and younger than 85 years old.
* BMI higher than 20 but lower than 40
* Patients with hypoxemia related to viral pneumonia (COVID-19) requiring oxygen or nasal high flow therapy (to maintain SpO2 above 92%) without criteria for immediate intubation or need for other respiratory supports (CPAP, non-invasive ventilation).
* Initiation of oxygen supplementation < 72 hours
* eGFR (CKD EPI) > 30 ml/min/1.73m2
* Serum troponin i < 80 ng/L
* Heart rate ≥ 55 bpm if beta blockers or calcium channel blocker nondihydropyridine are used, and ≥ 60 bpm in the other patients

Exclusion criteria Medical conditions

* Level of care B (unless patient agrees to intubation at study enrollment), C or D (patient admitted for palliative care; or physician is not committed to life-sustaining therapies)
* No SpO2 signal available (only if FreeO2 apparatus is used)
* Patient agitation (only if FreeO2 apparatus is used)
* Severe untreated sleep apnea
* History of or currently active primary or secondary immunodeficiency
* Recent (within the last 6 months) occurrence of myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, class III/IV heart failure
* Known presence of Mobitz type II second-degree or third-degree atrioventricular block, sick sinus syndrome, or sinoatrial block, unless patient has a functioning pacemaker
* Child-Pugh score class C
* Pregnancy, lactation, or a positive serum beta human chorionic gonadotropin measured during screening
* Persistent hypotension.

Prior/concomitant therapy

* Receipt of a live vaccine within 4 weeks prior to randomization
* Receiving MAO inhibitor (tranylcypromine, selegiline or phenelzine)
* Receiving pharmacological treatment for a form of multiple sclerosis
* Use of long-term immunosuppressors (Ex. tacrolimus, cyclosporin, azathioprine, mycophenolate, sirolimus, methotrexate or chronic use of corticosteroid (> 7.5 mg per day more than 3 months)
* Receiving Class Ia and class III anti-arrythmic drugs amiodarone, sotalol, flecainide, propafenone
* Patients receiving or anticipated to receive hydroxychloroquine or azithromycin.

Prior/concurrent clinical study experience -Current enrolment in an interventional arm of a clinical trial with similar endpoints to the COZI trial

Other exclusions

-Patients or legal/authorized representatives who refuse to participate to the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Daily Patient progression assessed with the World Health Organization-adapted 6-points ordinal scale | through whole duration of the hospitalization, an average of 14 days
  Clinical improvement until hospital discharge

SECONDARY OUTCOMES:
The mean oxygen flow required to maintain the oxygen saturation (SpO2) target at 92% | First 7 days of the trial
  Titrated every second with automated oxygen titration device (FreeO2)
Rate of non invasive ventilation (NIV) / high flow nasal therapy (HFNT) use | through whole duration of the hospitalization, an average of 14 days
Rate of intubation | through whole duration of the hospitalization, an average of 14 days
Ventilator-free and oxygen-free days at day 28 | through whole duration of the hospitalization, an average of 14 days
Rate of ICU admission/length of stay/mortality | through whole duration of the hospitalization, an average of 14 days
Severity index measurement | through whole duration of the hospitalization, an average of 14 days
  Sepsis-related organ failure assessment (SOFA), national early warning score (NEWS2), early warning score for oxygen therapy (EWS.O2), decrease of at least 2 points on the 6-point ordinal scale

CONTACTS AND LOCATIONS:
Overall Officials: François Lellouche, MD, Principal Investigator — IUCPQ-UL; David Marsolais, PhD, Study Chair — CRIUCPQ-UL; Nathalie Châteauvert, B. pharm, Study Chair — CRIUCPQ-UL; Pascale Blais-Lecours, PhD, Study Director — CRIUCPQ-UL
Locations (3):
- Canada (3):
  - Hôpital de la Cité-de-la-Santé (CISSS de Laval), Laval, Quebec
  - Hôpital Santa Cabrini Ospedale (CIUSSS EMTL), Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lellouche F, Blais-Lecours P, Maltais F, Sarrazin JF, Rola P, Nguyen T, Chateauvert N, Marsolais D. Ozanimod Therapy in Patients With COVID-19 Requiring Oxygen Support: A Randomized Open-Label Pilot Trial. Chest. 2024 Apr;165(4):810-819. doi: 10.1016/j.chest.2023.10.023. Epub 2023 Oct 28. PMID 37898184